CLINICAL TRIAL: NCT02247050
Title: Primary Care Clinician Commitments to Choosing Wisely®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Robert Wood Johnson Foundation (Other); IHA (Unknown)
Responsible Party: Principal Investigator, Jeffrey T. Kullgren, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00087820; 71475 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Health Services Misuse; Physician's Practice Patterns; Guideline Adherence; Unnecessary Procedures; Health Care Costs
Keywords: Costs and Cost Analysis; Professional Practice; Attitude of Health Personnel; Health Knowledge, Attitudes, and Practice; Decision Making; Practice Guidelines as Topic; Physician-Patient Relations; Physician's Role; Health Care; Quality of Health Care; Quality Assurance; Physicians, Primary Care; Evidence-Based Medicine; Evidence-Based Practice; Decision Support Systems, Clinical; Reminder Systems; Judgment; Cognition; Patient Care; Health Services Misuse; Unnecessary Procedures; Prescribing Patterns, Physician; Inappropriate Prescribing; Over Prescribing; Low Back Pain; Sinusitis; Infections, Upper Respiratory; Generalized Headache; Imaging, Diagnostic; Antibiotics; Humans; Overuse of Low-Value Services; Pragmatic Trial; Stepped Wedge Design; Cluster Randomized Trial; Choosing Wisely
MeSH Terms: conditions — Behavior; Low Back Pain; Sinusitis; Respiratory Tract Infections; Headache; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Commitment invitation at time 1 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the first clinic will remain in the control period (no intervention) for 2 months and then cross over to the intervention period for 6 months.
  Interventions: Behavioral: Commitment invitation
- Commitment invitation at time 2 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the second clinic will remain in the control period (no intervention) for 3 months and then cross over to the intervention period for 5 months.
  Interventions: Behavioral: Commitment invitation
- Commitment invitation at time 3 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the third clinic will remain in the control period (no intervention) for 4 months and then cross over to the intervention period for 4 months.
  Interventions: Behavioral: Commitment invitation
- Commitment invitation at time 4 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the fourth clinic will remain in the control period (no intervention) for 5 months and then cross over to the intervention period for 3 months.
  Interventions: Behavioral: Commitment invitation
- Commitment invitation at time 5 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the fifth clinic will remain in the control period (no intervention) for 6 months and then cross over to the intervention period for 2 months.
  Interventions: Behavioral: Commitment invitation
- Commitment invitation at time 6 (Experimental): Intervention: Behavioral: Commitment Invitation
  In the stepped wedge cluster randomized design, the sixth clinic will remain in the control period (no intervention) for 7 months and then cross over to the intervention period for 1 month.
  Interventions: Behavioral: Commitment invitation

INTERVENTIONS:
Behavioral: Commitment invitation — Clinicians will be invited to commit to follow 3 Choosing Wisely recommendations. Those that choose to commit will also receive point-of-care commitment reminders, point-of-care Choosing Wisely patient education handouts, and weekly emails with decision support resources.

SUMMARY:
This pragmatic trial examines the uptake and effects of primary care clinician commitments to follow 3 Choosing Wisely® recommendations. The investigators hypothesize that pre-encounter invitations to clinicians to commit to the recommendations will decrease ordering of: (1) imaging tests for low back pain, (2) antibiotics for acute sinusitis, and (3) imaging tests for headaches. The study is a mixed-methods, stepped wedge cluster randomized trial in which the intervention will be sequentially introduced to 6 clinics in southeastern Michigan in a randomly assigned order.

DETAILED DESCRIPTION:
Clinicians often make decisions about ordering low-value services in the midst of clinical encounters when their thinking can be rushed and susceptible to patient demands. This pragmatic trial examines the uptake and effects of shifting clinicians' decisions about ordering low-value services to the pre-encounter period when their thinking is slower and more deliberative; inviting clinicians to commit to avoid ordering those services during patient encounters; and providing to clinicians who committed decision support resources such as point-of-care reminders, patient education handouts, and access to brief communications training.

The investigators will conduct a mixed-methods, stepped wedge cluster randomized trial in 6 IHA primary care clinics in southeastern Michigan. The intervention will be introduced in each clinic in sequence approximately one month apart and in a randomly assigned order (i.e., temporal randomization). In each clinic the intervention will continue for 1 to 6 months so that the intervention ends in all clinics at the same time. For example, in the first clinic the intervention will run for 6 months; in the sixth clinic the intervention will run for 1 month. The total length of the control period plus the intervention period will be 8 months at all clinics.

Prior to the start of the study, IHA made its primary care clinicians aware of publicly available recommendations from the ABIM Foundation's Choosing Wisely® campaign applicable to avoiding overuse of low-value services for 3 common conditions: (1) low back pain, (2) acute sinusitis, and (3) headaches. However, research has shown that clinician behavior seldom changes as a result of information alone. Therefore, at the start of the intervention period clinicians will be invited to make a pre-encounter commitment to follow the 3 Choosing Wisely recommendations. Clinicians who choose to commit will throughout the intervention period receive point-of-care commitment reminders, Choosing Wisely patient education handouts, and weekly emails with decision support resources. Clinicians will remain free to order services at any time without penalty.

The investigators will measure whether the clinician-focused intervention leads to declines in rates of ordering imaging tests for low back pain, antibiotics for acute sinusitis, and imaging tests for headaches. The study team will analyze ordering patterns and costs using clinical operations datasets (drawn from electronic health records and from the billing and practice management system). The following hypotheses will be tested:

Hypothesis 1: Inviting primary care clinicians to commit to avoid ordering imaging for low back pain, antibiotics for acute sinusitis, and imaging for headaches will decrease ordering of these services.

Hypothesis 2: Inviting primary care clinicians to commit to avoid ordering imaging for low back pain, antibiotics for acute sinusitis, and imaging for headaches will reduce health care costs in patient visits for low back pain, acute sinusitis, and headaches.

Hypothesis 3: Inviting primary care clinicians to commit to avoid ordering low-value services will reduce per-clinician per-visit health care costs across clinical conditions.

For each outcome investigators will also compare differences between clinicians who did and did not commit to follow the 3 Choosing Wisely recommendations. Additionally, investigators will compare differences in outcomes between the 3-month follow-up period (immediately after the intervention has ended) and the control and intervention periods.

After the intervention period, the study team will conduct surveys and semi-structured interviews with study clinicians. The survey results will be used to identify correlates of primary care clinician uptake of invitations to commit to avoid ordering low-value services. The semi-structured interviews will elicit qualitative data on clinician attitudes towards overuse of low-value services, clinicians' responses to the intervention, and facilitators of and barriers to avoidance of delivering low-value care.

ELIGIBILITY:
Inclusion Criteria:

* Primary care clinicians in 6 primary care (family medicine and internal medicine) clinics within the IHA organization of Ann Arbor, Michigan

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite rates of ordering 3 potentially low-value services in primary care visits by adult patients | Within 10 months of receiving the intervention
  Composite rates of ordering lumbar spine imaging tests in visits for low back pain, ordering antibiotics in visits for acute sinusitis, and ordering head imaging tests in visits for headaches.

SECONDARY OUTCOMES:
Composite rates of ordering potential substitute services for 3 potentially low-value services in primary care visits by adult patients | Within 10 months of receiving the intervention
  Composite rates of ordering potential substitute services for lumbar spine imaging tests in visits for low back pain, ordering antibiotics in visits for acute sinusitis, and ordering head imaging tests in visits for headaches.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Kullgren, MD, MS, MPH, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - IHA Ann Arbor Family Medicine, Ann Arbor, Michigan
  - IHA Family Medicine - Arbor Park, Ann Arbor, Michigan
  - IHA Internal Medicine - Domino's Farms, Ann Arbor, Michigan
  - IHA Brighton Family Care, Brighton, Michigan
  - IHA Internal Medicine - Cherry Hill, Canton, Michigan
  - IHA Reichert Internal Medicine at Towsley, Ypsilanti, Michigan

REFERENCES:
- [Derived] Kullgren JT, Krupka E, Schachter A, Linden A, Miller J, Acharya Y, Alford J, Duffy R, Adler-Milstein J. Precommitting to choose wisely about low-value services: a stepped wedge cluster randomised trial. BMJ Qual Saf. 2018 May;27(5):355-364. doi: 10.1136/bmjqs-2017-006699. Epub 2017 Oct 24. PMID 29066616